CLINICAL TRIAL: NCT01355913
Title: Screening and Genetic Monitoring of Patients With MDS Under Different Treatment Modalities by Cytogenetic Analyses of Circulating CD34+Cells
Brief Title: Screening and Genetic Monitoring of Patients With Myelodysplastic Syndromes (MDS) Under Different Treatment Modalities by Cytogenetic Analyses of Circulating CD34+Cells
Status: Completed | Type: Observational
Sponsor: Institut fuer anwendungsorientierte Forschung und klinische Studien GmbH (Other)
Collaborators: University Medical Center Goettingen (Other)
Responsible Party: Detlef Haase, University Medical Center Goettingen
Other Study IDs: Diagnostik-Studie
Record Dates: First submitted 2011-05-17; First posted 2011-05-18 (Estimated); Last update posted 2020-02-21 (Actual); Status verified 2020-02

CONDITIONS: Myelodysplastic Syndromes (MDS); Chromosmal Aberrations; Karyotype Evolution; Rare Abnormalities; Cytogenetic Monitoring
Keywords: Myelodysplastic syndromes (MDS); chromosmal aberrations; cytogenetics; Fluorescence in situ hybridization (FISH); CD34+ cells; peripheral blood
MeSH Terms: conditions — Myelodysplastic Syndromes

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
In myelodysplastic syndromes (MDS) the knowledge about chromosomal aberrations is important for diagnosis, pathogenesis, prognosis and treatment. Usually, chromosomal anomalies in MDS patients are detected in bone marrow cells by chromosome banding analyses of metaphases. Alternatively or additionally they can be diagnosed by Fluorescence-in-Situ-Hybridization (FISH). The investigators here present a novel method for cytogenetic monitoring of MDS patients from peripheral blood which is representative for the clone size in bone marrow cells. The purpose of this prospective multicenter non-interventional diagnostic study is to detect and to follow chromosomal aberrations from peripheral blood closely, to assess karyotype evolution, to detect rare abnormalities and to correlate the molecular-cytogenetic results with peripheral blood counts, bone marrow morphology and treatment modalities and responses.

DETAILED DESCRIPTION:
Chromosomal aberrations in myelodysplastic syndromes (MDS) play a major role in diagnostics, pathogenesis, prognosis, and, more recently, in treatment allocations. Chromosomal anomalies can be detected by conventional chromosome banding analyses of bone marrow metaphases and most of them are provable by Fluorescence in situ hybridization (FISH) of circulating CD34+ progenitor cells from peripheral blood. For this prospective multicenter non-interventional diagnostic study sequential FISH analyses are performed on immunomagnetically enriched circulating CD34+ cells from peripheral blood as follows: A "super-panel" with the probes D7/CEP7, EGR1, CEP8, CEP XY, D20, p53, IGH/BCL2, TEL/AML1, RB1, MLL, 1p36/1q25, CSF1R (all Abbott® probes) is used for initial screening, every 12 months during follow-up and in every case of suspected progression. A smaller "standard-panel" with the probes EGR1, D7/CEP7, CEP8, p53, D20, CEP X/Y, TEL/AML1 - plus if necessary an informative probe of the superpanel- was performed for analyses at short intervals every 2 months in the 1st year and every 3 months during the 2nd and 3rd year. Peripheral blood counts are documented once a month, and full blood counts with the number of peripheral blasts are recommended at the time point of each FISH analysis. Bone marrow biopsies are not part of the study, but they are recommended to be performed every 6 to 12 months in the course of the disease. If a bone marrow biopsy is performed, conventional chromosome banding analyses on bone marrow metaphases and, additionally, FISH analyses of enriched CD34+ bone marrow cells and non-enriched bone marrow cells are performed. The results from peripheral blood are correlated with those of conventional banding and FISH analyses performed on bone marrow samples. The aims of this study are to detect acqired chromosomal aberrations in MDS patients from peripheral blood, to follow these anomalies by frequent analyses, to detect rare aberrations and to observe karyotype evolution from peripheral blood.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis (cytomorphologic proof) of primary or secondary myelodysplastic syndrome (MDS) or
* Suspected myelodysplastic syndrome (MDS).
* Age > 18 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 20 ml of peripheral blood (pb) of a MDS patient are enriched by immunomagnetic cell sorting (by MACS® system). A FISH analysis is performed on these CD34+ cells according to product protocols using the FISH probe panels described above. The percentage of aberrant interphase nuclei (IN) is measured related to all (at least 200) IN counted. FISH analyses are performed every 2 months in the 1st and every 3 months in the 2nd and 3rd year of follow-up by the same method using the standard panel and, if necessary, an informative probe of the super panel. Pb counts are documented once a month, and full blood counts with peripheral blasts are recommended at the time point of each FISH analysis. Bone marrow (bm) biopsies are not part of the study, but they are recommended to be performed every 6 to 12 months. If a bm biopsy is performed, conventional chromosome banding analyses on bm metaphases and FISH analyses of enriched CD34+ and non-enriched bm cells are performed.
Sampling Method: Probability Sample
Enrollment: 402 (Actual)
Dates: Start 2008-10 (Actual); Primary Completion 2016-10 (Actual); Study Completion 2019-10 (Actual)

PRIMARY OUTCOMES:
Screening and genetic monitoring of patients with MDS under different treatment modalities by cytogenetic analyses of circulating CD34+cells. | The first FISH analysis is performed at the time of study entry (initial screening) and after that every 2 months in the first year and every 3 months in the second and third year.
  At each timepoint of FISH analysis the percentage of aberrant interphase nuclei is measured of all (at least 200) interphase nuclei counted.

CONTACTS AND LOCATIONS:
Overall Officials: Detlef Haase, MD, Prof., Study Chair — University Medical Center Göttingen
Locations (13):
- Germany (13):
  - University Hospital Aachen, Aachen
  - University Hospital Dresden, Dresden
  - University Hospital Düsseldorf, Düsseldorf
  - Onkologikum, Frankfurt am Main
  - University Hospital Frankfurt/Main, Frankfurt am Main
  - Onkologische Kooperation Harz, Goslar
  - Group Practice Meyer/Ammon/Müller, Göttingen
  - University Medical Center Göttingen, Göttingen
  - Group Practice Uhle/Müller/Kröning/Jentsch-Ullrich, Magdeburg
  - Group Practice Schmidt/Galler/Klapthor, Munich
  - Technical University Munich, Munich
  - Group Practice Detken/Seraphin, Northeim
  - University Hospital Ulm, Ulm

REFERENCES:
- [Derived] Braulke F, Muller-Thomas C, Gotze K, Platzbecker U, Germing U, Hofmann WK, Giagounidis AA, Lubbert M, Greenberg PL, Bennett JM, Sole F, Slovak ML, Ohyashiki K, Le Beau MM, Tuchler H, Pfeilstocker M, Hildebrandt B, Aul C, Stauder R, Valent P, Fonatsch C, Bacher U, Trumper L, Haase D, Schanz J. Frequency of del(12p) is commonly underestimated in myelodysplastic syndromes: Results from a German diagnostic study in comparison with an international control group. Genes Chromosomes Cancer. 2015 Dec;54(12):809-17. doi: 10.1002/gcc.22292. Epub 2015 Sep 10. PMID 26355708
- [Derived] Braulke F, Platzbecker U, Muller-Thomas C, Gotze K, Germing U, Brummendorf TH, Nolte F, Hofmann WK, Giagounidis AA, Lubbert M, Greenberg PL, Bennett JM, Sole F, Mallo M, Slovak ML, Ohyashiki K, Le Beau MM, Tuchler H, Pfeilstocker M, Nosslinger T, Hildebrandt B, Shirneshan K, Aul C, Stauder R, Sperr WR, Valent P, Fonatsch C, Trumper L, Haase D, Schanz J. Validation of cytogenetic risk groups according to International Prognostic Scoring Systems by peripheral blood CD34+FISH: results from a German diagnostic study in comparison with an international control group. Haematologica. 2015 Feb;100(2):205-13. doi: 10.3324/haematol.2014.110452. Epub 2014 Oct 24. PMID 25344522
- [Derived] Braulke F, Jung K, Schanz J, Gotze K, Muller-Thomas C, Platzbecker U, Germing U, Brummendorf TH, Bug G, Ottmann O, Giagounidis AA, Stadler M, Hofmann WK, Schafhausen P, Lubbert M, Schlenk RF, Blau IW, Ganster C, Pfeiffer S, Shirneshan K, Metz M, Detken S, Seraphin J, Jentsch-Ullrich K, Bohme A, Schmidt B, Trumper L, Haase D. Molecular cytogenetic monitoring from CD34+ peripheral blood cells in myelodysplastic syndromes: first results from a prospective multicenter German diagnostic study. Leuk Res. 2013 Aug;37(8):900-6. doi: 10.1016/j.leukres.2013.03.019. Epub 2013 Apr 25. PMID 23623559